CLINICAL TRIAL: NCT06803628
Title: Contribution of Point of Care Ultrasound by the Emergency Physician to Rule Out the Small Bowel Obstruction: a Diagnostic, Multicenter Study
Acronym: OCCLUS-POCUS
Status: Recruiting | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC24_0388
Record Dates: First submitted 2025-01-27; First posted 2025-01-31 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Small Bowel Obstruction
Keywords: Small bowel obstruction; Point of care ultrasound; Emergency Medicine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- POCUS: Point of care ultrasound in Small bowel obstruction in Emergency Medicine,
  Interventions: Other: Point of care ultrasound

INTERVENTIONS:
Other: Point of care ultrasound — OCCLUS-POCUS will include patients with suspected SBO, with low or moderate Gestalt probability who meet the inclusion criteria During the patient's visit to the ED, the investigating physician will present the study and the importance of evaluating the value of POCUS in the diagnosis of exclusion of SBO. Once oral non-opposition to the study has been obtained, the participation of the patient lasts 28 days.
  POCUS is performed only for patients with low or moderate Gestalt probability. It will be performed by trained emergency physicians (EP) using a curvilinear probe . After POCUS realization, the EP will:
  * determine if there is presence or absence of SBO.
  * collect POCUS duration, difficulty and investigator's characteristics.
  * Realization of CT which will be the gold standard for SBO presence or absence.
  * The study protocol procedure ends when the report of the CT is available and the physician establish its diagnosis.
  * The study ends at D28 with a phone call

SUMMARY:
Small Bowel Obstruction (SBO) is a frequent pathology in the emergency department (ED). Diagnosis is currently based on abdominal CT scan (CT). Moreover, CT is warranted to determine the therapeutic strategy in patients with SBO which could include medical treatment; surgical intervention or both. However, CT is associated with drawbacks such as radiation exposure, increased cost and ED length-of-stay.

In a prospective observational study, a SBO was excluded by CT in 45% [95%CI: 37-53] of patients. There is, thus, a need for improving the appropriateness of CT-scan for suspected SBO.

A recent meta-analysis showed that Point of care ultrasound (POCUS) had a good diagnostic accuracy (sensitivity 83% [95%CI 71.7%-90.4%]), specificity 93% [95%CI 55.3%-99.3%]). Another meta-analysis found rather similar results (sensitivity 83% [(95% CI 89.0% to 94.7%], specificity 96,6% [95% CI 88.4% to 99.1%]).

In order to improve the negative predictive value of POCUS for its implementation as a rule-out strategy, CHU of Nantes emergency unit studied the combination of POCUS with Gestalt pre-test probability of SBO determined by the emergency physician. This SBO probability classified the patients as low, moderate or high risk of SBO. In patients with low or moderate Gestalt probability, CHU of Nantes emergency unit found that this combined strategy had a sensitivity of 100% [95% CI: 88-100] and NPV 100% [92-100%].

By (i) focusing on patients with a low or moderate Gestalt clinical probability and (ii) increasing the number of patients included, CHU of Nantes emergency unit intends to demonstrate that POCUS is able to exclude SBO in this population. This would avoid unnecessary CT and thus lower costs, ED length-of-stay and hospital radiologists workload.

A POCUS will be performed followed by a CT (gold standard). The main objective will be the ability of POCUS to rule-out SBO in patients with low or moderate Gestalt clinical probability.

DETAILED DESCRIPTION:
Small Bowel Obstruction (SBO) is a frequent pathology, leading to admissions to emergency departments (ED). Diagnosis is currently based on an abdominal CT scan (CT). However, CT is associated with drawbacks such as radiation exposure, increased cost and ED length-of-stay.

A recent meta-analysis including 1178 patients showed that Point of care ultrasound (POCUS) had a good diagnostic accuracy (sensitivity 83% [95%CI 71.7%-90.4%]), specificity 93% [95%CI 55.3% -99.3%]). Another meta-analysis with 433 patients, found rather similar results: sensitivity 83% [95% CI 89.0% to 94.7%], specificity 96,6% [95% CI 88.4% to 99.1%]).

Since CT is almost warranted to guide the treatment strategy, which could include surgery, medical treatment or both, CHU of Nantes emergency unit explored a different approach focusing on POCUS rule-out ability. This study also introduced the notion of SBO Gestalt probability which is a global clinical evaluation by the physician. Gestalt probability has mainly been explored in patients with suspected pulmonary embolism and was found as effective as clinical prediction rules. It is used in the routine clinical evaluation of patient with suspicion of pulmonary embolism. When applied to patients with SBO suspicion, the physician chooses between low, moderate or high risk of SBO. Based on CT results, prevalence of SBO based on Gestalt probability were 21%, 45% and 87% in the low, moderate and high risks, respectively.

Our team studied POCUS with the following items that were searched in the whole abdomen divided into nine zones: dilated incompressible fluid-filled intestinal loop (>25 mm) with back-and-forth fluid movement. When at least one of these signs was present in one zone, the SBO was highly suspected. As it was an observational study, a CT was performed in all patients and was the gold standard. This approach was associated with a POCUS sensitivity in the whole population of 99% [95% CI: 93-99.8] [2]. POCUS would thus have a role in patients with low and moderate SBO risks because the prevalence of SBO was major in the high risk Gestalt probability category of patients, and thus CT is the only imaging needed in these latter. Furthermore, in patients with low or moderate probability, the sensitivity was 100% [95% CI: 88-100] In previous studies, the sensitivity was not able to exclude SBO with sufficient security since the lower 95% confidence interval margin was near 90%. By (i) focusing on patients with a low or moderate clinical Gestalt probability and (ii) increasing the number of patients, CHU of Nantes emergency unit intends to demonstrate that POCUS should be able to safely exclude SBO in this population.

In case of positive results, the diagnostic strategy in case of SBO suspicion could be modified in: firstly, assess the clinical Gestalt probability; secondly perform a POCUS in patients with low or moderate Gestalt probability and thirdly, prescribe a CT only for patients with high clinical probability or presence of POCUS signs of SBO. This would avoid unnecessary CT and thus lower patient's.

exposure, costs, ED length-of-stay and radiologist workload. A study performed in the USA simulated a POCUS first approach in patients with suspected SBO and found that it could save ED length of stay, radiation and money. In France in 2017, about ¾ of ED were equipped with ultrasound machines and half of the emergency physicians were trained in POCUS. Furthermore, SBO detection is easily performed: in our study, the operator self-assessed ultrasound experience was beginner or intermediate for 59% of patients. In case of positive results, this technique would be largely deployed.

Inclusion criteria will be patients with low or moderate Gestalt clinical probability of SBO. A POCUS will be performed followed by a CT (gold standard). This CT will be realized and interpreted blindly from the POCUS results. The main objective will be the ability of POCUS to rule-out SBO in patients with low or moderate Gestalt clinical probability

ELIGIBILITY:
Inclusion Criteria:

1. Major patient (age > 18 years old), no upper limit
2. Patient admitted to the ED with suspected SBO (abdominal pain, vomiting, cessation of gas and feces...)
3. Low or moderate pretest Gestalt clinical probability
4. Patient able to understand protocol and express agreement
5. Oral non-opposition given

Exclusion Criteria:

1. Patient under legal guardianship
2. Pregnant women
3. Nursing mothers
4. Patient who does not speak or understand French
5. Patient without a health insurance plan
6. Patient who already had imaging confirming the diagnosis
7. Patient who participates simultaneously in any interventional study focused on abdominal pain before POCUS and CT realization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with suspected SBO, with low or moderate Gestalt probability and who meet the inclusion criteria (and without any non inclusion criteria)
Sampling Method: Non-Probability Sample
Enrollment: 667 (Estimated)
Dates: Start 2025-03-10 (Actual); Primary Completion 2027-03-10 (Estimated); Study Completion 2027-03-10 (Estimated)

PRIMARY OUTCOMES:
Estimate the ability of POCUS to rule-out SBO in patients with low or moderate Gestalt clinical probability | Day 1
  Evaluation of the negative predictive value (NPV) of point of care ultrasound (POCUS) in patients with suspected Small Bowel Obstruction (SBO) (number of patients with negative POCUS in patients without SBO according to the CT (gold standard) divided by total patients with negative POCUS)

SECONDARY OUTCOMES:
1/ Diagnostic accuracy of POCUS for the diagnosis of SBO | Day 1
  1/ Sensitivity, specificity, positive predictive value of POCUS determined from POCUS and CT results.
2/ Estimation of time between POCUS and CT report | Day 1
  2/ Time between point of care ultrasound and CT report
3a/ Description of "false negative" (exclusion of SBO diagnosis by POCUS, but diagnosis of SBO by CT) | Day 1
  3a/ Characteristics associated with false negative (BMI, sex, age, physician's experience, physician's evaluation of POCUS difficulty on a numerical scale from 0 to 10)
3b/ Description of "false positive" (SBO diagnosis by POCUS, but diagnosis of SBO excluded by CT) | Day 1
  3b/ Characteristics associated with false positive (BMI, sex, age, physician's experience, physician's evaluation of POCUS difficulty on a numerical scale from 0 to 10)
4/ Description of patients with a final diagnosis other than SBO | Day 1
  4/ Patients' characteristics with other diagnosis than SBO (BMI, sex, age, final diagnosis)
5/ Physician's assessment of the POCUS procedure | Day 1
  5/ Duration in minutes of POCUS and difficulty of clinical POCUS estimated by the operator on a numerical scale named "operator difficulty of clinical POCUS realization" from 0 to 10 (0 being the lower and 10 the higher score)
6a/ Physician intention to prescribe CT even if POCUS showed no SBO | Day 1
  6a/ Number of CT which would have been prescribed for acute abdominal pain
6b/ Reason for which CT would have been realized | Day 1
  6b/ Reason for requesting a CT in spite of exclusion of a diagnosis of SBO (poor echogenicity, lack of confidence in its realization, other diagnostic suspicion requiring a CT scan …)
7/ Follow-up of patients | Day 28
  Phone call at Day 28 to establish the health status in relation to the previous reason for emergency consultation, to know if a second visit to emergency department for same reason within 7 days of primary consultation happened, and/or if another hospitalization within 28 days happened)

CONTACTS AND LOCATIONS:
Locations (18):
- France (18):
  - Chu Clermont-Ferrand Hopital Gabriel Montpied, Clermont-Ferrand, France
  - Ghem Groupe Hospitalier Eaubonne Montmorency Simone Veil, Eaubonne, France
  - CHD Vendée, La Roche-sur-Yon, France
  - CHD Vendée, Luçon, Luçon, France
  - Ap-Hm Hopital La Timone, Marseille, France
  - Hôpital Nord, Marseille, France
  - Ghsif Groupe Hospitalier Sud Ile de Franc _ Ch Melun, Melun, France
  - CHD Vendée, Montaigu, Montaigu, France
  - CHU Nantes, Nantes, France
  - Le Confluent, Nantes, France
  - CHU CAREMEAU - Nimes, Nîmes, France
  - AP-HP Est Parisien _ ST-ANTOINE, Paris, France
  - P-HP Paris Centre - COCHIN, Paris, France
  - Chru Poitiers, Poitiers, France
  - CH MEMORIAL - Saint Lô, Saint-Lô, France
  - CH Saint-Nazaire, Saint-Nazaire, France
  - Groupe Hospitalier Selestat Obernai (Ghso), Sélestat, France
  - Hopital PURPAN CHU Toulouse, Toulouse, France

IPD SHARING:
Plan to Share IPD: No